CLINICAL TRIAL: NCT02793895
Title: Post-Surgical Enhanced Monitoring for Cardiac Arrhythmias and Atrial Fibrillation (SEARCH-AF): A Randomized Controlled Trial
Brief Title: Detection of Atrial Fibrillation After Cardiac Surgery
Acronym: SEARCH-AF
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 pandemic
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: SEARCH-AF-001; NCT04145648 (obsolete NCT alias)
Record Dates: First submitted 2016-05-02; First posted 2016-06-08 (Estimated); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Atrial Fibrillation; Atrial Flutter; C.Surgical Procedure; Cardiac; Arrhythmias, Cardiac
Keywords: Atrial fibrillation/flutter; Postoperative atrial arrhythmia; Cardiac surgery; Stroke prevention; Oral anticoagulation; Cardiac rhythm monitoring
MeSH Terms: conditions — Atrial Fibrillation; Atrial Flutter; Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced cardiac rhythm monitoring (Experimental): Subjects in this group will receive up to 30 days of continuous cardiac rhythm monitoring with an adhesive monitor. Cardiac rhythm monitoring will begin on the day of randomization. The device that will be used is the Medtronic SEEQ™ mobile cardiac telemetry system or the CardioSTAT (Icentia Inc.) cardiac rhythm monitoring device. At 6+/-1 months, subjects randomized to the intervention group will undergo 14 days of continuous cardiac rhythm monitoring with the SEEQ™ device or the CardioSTAT (Icentia Inc.) cardiac rhythm monitoring device.
  Interventions: Device: Medtronic SEEQ™ mobile cardiac telemetry system; Device: CardioSTAT (Icentia Inc.) cardiac rhythm monitoring device
- Usual care (Active Comparator): Subjects randomized to the usual care arm will be discharged from hospital without protocol-mandated continuous cardiac rhythm monitoring. Within the first 30 days after randomization, no protocol-mandated cardiac rhythm assessment will be arranged. At 6+/-1 months, subjects randomized to the usual care group will undergo 14 days of continuous cardiac rhythm monitoring with the SEEQ™ device or the CardioSTAT (Icentia Inc.) cardiac rhythm monitoring device.
  Interventions: Other: Usual Care

INTERVENTIONS:
Device: Medtronic SEEQ™ mobile cardiac telemetry system — The SEEQ™ system consists of a wearable sensor which is a single-lead, low-profile, peel-and-stick device applied over the anterior left chest wall of the subject. The wearable patch is designed for one-time use only and cannot be re-applied if removed. Each sensor provides up to 7.5 days of monitoring. Subjects randomized to the intervention group will undergo 30 days of continuous cardiac rhythm monitoring with the SEEQ™ device at the time of randomization. At 6+/-1 months, subjects randomized to the intervention group will undergo 14 days of continuous cardiac rhythm monitoring with the SEEQ™ device.
  Arms: Enhanced cardiac rhythm monitoring
Other: Usual Care — For subjects randomized to the usual care group, no protocol-mandated cardiac rhythm monitoring will be performed. However, subjects in the control group may undergo rhythm monitoring during the study period if their treating physicians deem that there is a clinical indication to so do. At 6+/-1 months, subjects randomized to the usual care group will undergo 14 days of continuous cardiac rhythm monitoring with the SEEQ™ device or the CardioSTAT (Icentia. Inc) cardiac rhythm monitoring device.
  Arms: Usual care
Device: CardioSTAT (Icentia Inc.) cardiac rhythm monitoring device — The CardioSTAT device is a wearable adhesive cardiac rhythm monitoring system which is low-profile, water-resistant, and is adhered onto the skin surface with 2 electrodes. This wearable adhesive device is designed for one-time use only. Each CardioSTAT device will provide 14 days of cardiac rhythm monitoring. For subjects randomized to the intervention group who will be monitored by the CardioSTAT device, they will receive 28 days of continuous cardiac rhythm monitoring.
  Arms: Enhanced cardiac rhythm monitoring

SUMMARY:
The aim of the SEARCH-AF trial is to evaluate a novel diagnostic tool for detecting post-operative atrial fibrillation or flutter (POAF/AFL) in cardiac surgical subjects during the early, sub-acute post-operative period. The population includes cardiac surgical subjects who have either developed or are at risk for developing new onset POAF/AFL and who are at risk for stroke, as determined by their CHA2DS2-VASC (congestive heart failure, hypertension, age ≥75 years (2 points), diabetes mellitus, previous stroke/transient ischemic attack (TIA) (2 points), vascular disease, age 65-74 years, sex class (female)) score. These subjects must not have had a history of AF/AFL before cardiac surgery.

The intervention group will undergo up to 30 days of continuous cardiac rhythm monitoring with an adhesive, patch-based monitor (Medtronic SEEQ™ mobile cardiac telemetry system or the CardioSTAT (Icentia Inc.) cardiac rhythm monitoring device). The control group will receive usual care, which does not involve planned cardiac rhythm testing within the first 30 days after study randomization. The primary outcome is documentation of sustained atrial fibrillation or flutter within the first 30 days after randomization. In addition, subjects in both groups will undergo 14 days of continuous cardiac rhythm monitoring with the Medtronic SEEQ™ mobile cardiac telemetry system or the CardioSTAT (Icentia Inc.) cardiac rhythm monitoring device at 6±1 months after their index cardiac surgery.

DETAILED DESCRIPTION:
The aim of the SEARCH-AF trial is to evaluate a novel diagnostic tool for detecting post-operative atrial fibrillation or flutter (POAF/AFL) in cardiac surgical subjects during the early, sub-acute post-operative period. Its primary objective is to test whether enhanced cardiac rhythm monitoring with an adhesive, continuous monitor results in higher rates of atrial fibrillation or flutter (AF/AFL) detection at 30 days after randomization for post-cardiac surgical subjects who are at risk for developing post-operative atrial arrhythmias, when compared to usual care.

The study design is an open-label, two-arm randomized controlled trial (RCT) comparing a strategy of enhanced cardiac rhythm monitoring vs. usual care in 396 post-cardiac surgical subjects who are at risk for developing POAF/AFL.

The primary endpoint is the proportion of subjects with a cumulative AF/AFL burden of ≥6 minutes or documentation of AF/AFL by a 12-lead ECG within 30 days after randomization. Clinical endpoints will be adjudicated by an independent committee of physicians.

The study population involves post-cardiac surgical subjects at high risk of stroke, defined as having a CHA2DS2-VASC score of ≥4 or CHA2DS2-VASC of ≥2 with additional risk factors for developing POAF/AFL. These subjects must not have a history of AF/AFL pre-operatively.

Subjects who meet inclusion criteria will be randomized in a 1:1 ratio to one of the following 2 arms: (i) Enhanced cardiac rhythm monitoring (intervention group) or (ii) Usual care (control group). Subjects in the intervention group will receive up to 30 days of continuous cardiac rhythm monitoring with the Medtronic SEEQ™ mobile cardiac telemetry system or the CardioSTAT (Icentia Inc.) cardiac rhythm monitoring device. Monitoring will begin on the day of randomization. Subjects in the usual care group will not undergo protocol-mandated cardiac rhythm monitoring during the first 30 days after randomization.

All subjects will have a follow-up visit at 31-90 days after hospital discharge and at 6±1 months after surgery. At 6±1 months, all subjects will undergo 14 days of continuous cardiac rhythm monitoring with the SEEQ™ mobile cardiac telemetry system or the CardioSTAT (Icentia Inc.) cardiac rhythm monitoring device. A telephone follow-up will be performed for all subjects at 9±1 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female age ≥18 years.
2. Isolated CABG or valve replacement/repair +/- CABG performed at the index surgical procedure.
3. At elevated risk of stroke and for having POAF/AFL, defined as having a CHA2DS2-VASC (congestive heart failure, hypertension, age ≥75 years (2 points), diabetes mellitus, previous stroke/transient ischemic attack (TIA) (2 points), vascular disease, age 65-74 years, sex class (female)) score of ≥4 or ≥2 with at least 1 of the following risk factors for developing POAF/AFL:

   (i) Chronic obstructive pulmonary disease; (ii) Sleep apnea; (iii) Impaired renal function (defined as creatinine clearance <60 ml/min/1.73m2 or <60 ml/min); (iv) Echocardiographic evidence of at least mild left atrial enlargement (defined as ≥41 mm on M-mode, ≥59 ml or ≥29 mL/m2 on biplane volume assessment from an echocardiogram performed within 12 months of study enrollment); (v) Elevated body mass index (defined as BMI ≥30); (vi) Combined surgery (CABG + valve repair/replacement).
4. Able to provide written informed consent.

Exclusion Criteria:

1. Atrial fibrillation or flutter at the time of randomization.
2. Known previous history of AF/AFL, diagnosed pre-operatively (note: documentation of a history of AF/AFL without accompanying rhythm proof will suffice).
3. Documentation of continuous AF/AFL for ≥24 hours during the in-hospital stay for the index cardiac surgery.
4. Subjects who, at the discretion of the treating cardiac surgery team, would be treated and discharged with oral anticoagulation due to POAF/AFL.
5. Mechanical valve replacement.
6. Current or anticipated treatment with oral anticoagulation for indications other than AF/AFL.
7. Hospitalization for ≥10 days (for the index cardiac surgery, with day #0 being the day of surgery).
8. Planned discharge from hospital with a type IC or III anti-arrhythmic drug.
9. Having received >5 grams of IV and/or oral amiodarone during hospitalization for the index cardiac surgical procedure.
10. Women of childbearing potential (WOCBP).
11. History of percutaneous or surgical left atrial ablation for AF.
12. Presence of a cardiac implantable electronic device with a functioning atrial lead (pacemaker, implantable cardioverter defibrillator, or cardiac resynchronization device).
13. Presence of an implantable loop recorder.
14. History of left atrial appendage ligation, removal, or occlusion.
15. Subjects with known allergies or hypersensitivities to adhesives or hydrogel.
16. Inability to provide written informed consent.
17. Current or anticipated participation in another randomized controlled trial in which the interventional drug or device is known to affect the incidence of the primary or secondary outcomes of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 336 (Actual)
Dates: Start 2017-02-24 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-09-11 (Actual)

PRIMARY OUTCOMES:
Number of participants with a cumulative atrial fibrillation/flutter (AF/AFL) duration of ≥6 minutes or documentation of AF/AFL by a 12-lead electrocardiogram | Within 30 days of randomization.
  The primary endpoint of this trial is documentation of sustained AF/AFL, defined as a cumulative AF/AFL duration of ≥6 minutes or documentation of AF/AFL by a 12-lead ECG within 30 days after randomization. Clinical endpoints will be adjudicated by an independent clinical events committee.

SECONDARY OUTCOMES:
Number of participants with atrial fibrillation or flutter lasting for ≥24 hours. | (i) Within 30 days of randomization and (ii) Between day 31 and the last follow-up date.
  This outcome will be measured by a continuous cardiac modality (e.g. Holter, Event monitor, SEEQ™ mobile cardiac telemetry system, CardioSTAT (Icentia Inc.) cardiac rhythm monitoring device).
Duration of cumulative atrial fibrillation or flutter burden amongst participants. | Between day 31 of randomization and the last follow-up date.
  This outcome will be measured by a continuous cardiac modality (e.g. Holter, Event monitor, SEEQ™ mobile cardiac telemetry system, CardioSTAT (Icentia Inc.) cardiac rhythm monitoring device).
Number of participants who are prescribed with oral anticoagulation for atrial fibrillation or flutter-related stroke prevention. | (i) Within the first 45 days after discharge from cardiac surgery; (ii) Between day 46 and the last follow-up date.
  This outcome will be collected during study follow-up visits.
Number of days during which the adhesive Medtronic SEEQ™ or CardioSTAT (Icentia Inc.) cardiac rhythm monitoring device was worn by participants. | (i) Within 30 days after randomization (intervention group only); (ii) Between day 31 and the last follow-up date (all subjects).
  This outcome will be collected during study follow-up visits.
Number of participants who prematurely remove the adhesive Medtronic SEEQ™ or CardioSTAT (Icentia Inc.) cardiac rhythm monitoring device. | (i) Within 30 days after randomization (intervention group only); (ii) Between day 31 and the last follow-up date (all subjects).
  This outcome will be collected during study follow-up visits.
Number of participants with adverse events related to the use of the Medtronic SEEQ™ or CardioSTAT (Icentia Inc.) cardiac rhythm monitoring device. | (i) Within 30 days after randomization (intervention group only); (ii) Between day 31 and the last follow-up date (all subjects).
  This outcome will be collected during study follow-up visits.
Number of participants who undergo non-protocol mandated Holter monitoring and/or event recorders. | (i) Within 30 days after randomization; (ii) Between day 31 and the last follow-up date.
  This outcome will be collected during study follow-up visits.
Hospitalization or emergency room visits. | Within the first 45 days after hospital discharge from index cardiac surgery.
  This outcome will be collected during study follow-up visits.
Major adverse cardiac outcomes. | (i) Within the first 45 days after hospital discharge from index cardiac surgery; (ii) Between day 46 and the last follow-up date.
  All-cause death, myocardial infarction, ischemic stroke, non-CNS systemic embolism.
Number of participants with bleeding events. | (i) Within the first 45 days after hospital discharge from index cardiac surgery; (ii) Between day 46 and the last follow-up date.
  Major bleeding.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew CT Ha, MD, Principal Investigator — University Health Network, Toronto; Atul Verma, MD, Principal Investigator — St. Michael's Hospital and Southlake Regional Health Centre; Subodh Verma, MD, PhD, Principal Investigator — Unity Health Toronto
Locations (10):
- Canada (10):
  - St. Boniface General Hospital, Winnipeg, Manitoba
  - Saint John Regional Hospital, Saint John, New Brunswick
  - Kingston General Hospital, Kingston, Ontario
  - Southlake Regional Health Centre, Newmarket, Ontario
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - University Health Network, Toronto, Ontario
  - Université Laval, Québec, Quebec
  - Foothills Medical Centre, Calgary
  - Mazankowski Alberta Heart Institute, Edmonton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ha ACT, Verma S, Mazer CD, Quan A, Yanagawa B, Latter DA, Yau TM, Jacques F, Brown CD, Singal RK, Yamashita MH, Saha T, Teoh KH, Lam BK, Deyell MW, Wilson M, Hibino M, Cheung CC, Kosmopoulos A, Garg V, Brodutch S, Teoh H, Zuo F, Thorpe KE, Juni P, Bhatt DL, Verma A; SEARCH AF CardioLink-1 Investigators. Effect of Continuous Electrocardiogram Monitoring on Detection of Undiagnosed Atrial Fibrillation After Hospitalization for Cardiac Surgery: A Randomized Clinical Trial. JAMA Netw Open. 2021 Aug 2;4(8):e2121867. doi: 10.1001/jamanetworkopen.2021.21867. PMID 34448866
- [Derived] Yanagawa B, Ad N, Gaudino MF. Commentary: Postoperative atrial fibrillation can last years? Oh snap! J Thorac Cardiovasc Surg. 2020 Apr;159(4):1417-1418. doi: 10.1016/j.jtcvs.2019.04.028. Epub 2019 Apr 24. No abstract available. PMID 31155412